CLINICAL TRIAL: NCT02700906
Title: Corticosteroid and Lidocain Injections for Tennis Elbow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Principal Investigator, Lin-Fen Hsieh, Chief, Shin Kong Wu Ho-Su Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20130713R
Record Dates: First submitted 2016-02-02; First posted 2016-03-07 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-03

CONDITIONS: Tennis Elbow; Lateral Epicondylitis
Keywords: Lateral epicondylitis; tennis elbow; Lidocaine; corticosteroid
MeSH Terms: conditions — Tennis Elbow | interventions — Adrenal Cortex Hormones; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Corticosteroid injection (Active Comparator): For corticosteroid injection, triamcinolone (10mg/ml) 1 ml will be injected to the lateral epicondyle of the affected elbow.
  Interventions: Drug: Corticosteroid
- Lidocaine injection (Active Comparator): For lidocain injection, 1ml 1% lidocain will also be peppered on the same area.
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Corticosteroid — triamcinolone (10mg/ml) 1 ml will be injected to the lateral epicondyle of the affected elbow.
  Arms: Corticosteroid injection
Drug: Lidocaine — For lidocain injection, 1ml 1% lidocain will also be peppered on the same area.
  Arms: Lidocaine injection

SUMMARY:
The investigators hypothesized that lidocain injection is as effective as corticosteroid injection in management of tennis elbow, and if so, it may replace corticosteroid injection in the management of tennis elbow.

DETAILED DESCRIPTION:
Lateral epicondylitis or tennis elbow is a tendinopathy of the common extensor origin of the lateral elbow, and is estimated to have an annual incidence of 1-3%. It is characterized by tenderness over the lateral epicondyle of the humerus, normal range of motion, and pain on resisted extension of the wrist or fingers. Symptoms can persist for between 6 months and 2 years but usually resolve within 12 months. Although tennis elbow is often self-limited, around 20% of cases are refractory to conservative care. Tennis elbow is now thought to be non-inflammatory, and the pathologies are characterized by collagen degeneration, fibroblast proliferation, mucoid degeneration, and neovascularization.

Treatment of tennis elbow includes relative rest, physical therapy (therapeutic exercise, massage, therapeutic ultrasound, lower power laser, etc.), analgesics, non-steroidal anti-inflammatory drugs, glyceryl trinitrate patches, injection therapy (corticosteroid, hyaluronan gel, botulinum toxin, and autologous platelet-rich plasma), shock wave therapy, and even surgery. Previous studies showed corticosteroid injection is effective in the short term, but is harmful in the long-term, and is more likely to have a recurrence. In consideration of a degenerative lesion in tennis elbow, corticosteroid injection may be not an ideal agent. Although plate-rich plasma injection showed promising results, the high cost limited its widespread clinical use. Since local lidocain injection is commonly used in the management of myofascial pain syndrome, it might be effective in the treatment of tendinopathy like tennis elbow. The purpose of this study is to compare the effect of corticosteroid injection and lidocain injection in the treatment of tennis elbow. The investigators hypothesized that lidocain injection is as effective as corticosteroid injection in management of tennis elbow, and if so, it may replace corticosteroid injection in the management of tennis elbow.

ELIGIBILITY:
Inclusion Criteria:

* Between 20 and 75 years of age, with lateral elbow pain ≥4 in pain VAS for at least 1 month
* Reproducibility of pain by 2 or more of the following tests: palpation of the lateral epicondyle and/or the common extensor origin of the elbow; resisted wrist extension (dorsiflexion) and pronation with the elbow in extension
* Pain reproduced by static stretching of the pronated wrist in palmar flexion with the elbow in extension.

Exclusion Criteria:

* not fulfill inclusion criteria

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
change in the composite score on the Patient-Rated Tennis Elbow Evaluation (PRTEE) | baseline, 2 weeks, 2 months
  The primary outcome measure is the change in the composite score on the Patient-Rated Tennis Elbow Evaluation (PRTEE), which is a tennis elbow-specific questionnaire evaluating disease-specific quality of life. PRTEE includes a 5-item pain scale, with o indicating no pain and 10 indicating the worst pain imaginable; a 10-item functional disability scale, with 0 indicating no difficulty and 10 indicating greatest difficulty (unable to do). The scores range from 0 (good quality-of- life, no pain or disability) to 100 (poor-quality of-life, extremes pain and disability).

SECONDARY OUTCOMES:
pain-free grip strength | baseline, 2 weeks, 2 months
  The grip strength is a commonly used objective measure of tennis elbow-related disability, with good test-retest (Pearson correlation, r≥0.80) and validity (±3%) measures. The participants will sit in a chair with their shoulder flexed at 90 degrees, their elbows extended, and their forearms in neutral position. All participants are instructed to squeeze the dynamometer and cease squeezing before the onset of pain. The mean of the three replications will be recorded, with each measure separated by 60-sec interval.
ultrasound elbow assessment | baseline, 2 weeks, 2 months
  Another secondary outcome measure is ultrasound assessments of common extensor tendons at elbow, using published ordinary scales for hypoechogenecity, tendon thickness, and neovascularity, which have been reported to be associated tendinopathy.
treatment satisfaction | baseline, 2 weeks, 2 months
  Treatment satisfaction included patient's rating of the treatment outcome, using a 5-point(0, very dissatisfied; 5 very satisfied) scale.

CONTACTS AND LOCATIONS:
Overall Officials: Lin-Fen Lin-Fen, M.D, Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No